CLINICAL TRIAL: NCT01776450
Title: Compassionate Use of the Incraft® AAA Stent Graft System
Status: No longer available | Type: Expanded Access
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: G120003/S4
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

INTERVENTIONS:
Device: Endovascular AAA repair

SUMMARY:
To treat patients with abdominal aortic aneurysms requiring endovascular repair outside of the clinical protocol through compassionate use.

DETAILED DESCRIPTION:
In the US, abdominal aortic aneurysms (AAA) are found in 4-8% of older men and 0.5-1.5% of older women, resulting in 30,000-40,000 elective procedures and 1,400 peri-operative deaths. The most significant complication of AAA is an aneurysm sac rupture from which more than 15,000 patients die annually and is the 15th leading cause of death in elderly between 60 to 85 years of age . In Japan, it is estimated that approximately 14,000 endovascular aneurysm repair (EVAR) and open surgical repair cases were performed in the year 2010 .

Abdominal aortic aneurysms can be treated three ways: (1) Medical management; (2) Open surgical repair; and (3) Endovascular aneurysm repair (EVAR). EVAR has emerged as an alternative treatment of AAA for most patients. It is less invasive than open repair and carries lower rates of early mortality and morbidity . It has also extended treatment options to patients who cannot undergo conventional surgical procedures due to a high operative risk. As EVAR technology evolves, it allows treatment of AAA with increasing complexity of the aortic neck and access vessels.

The InCraft ®AAA Stent Graft System is designed for endovascular repair of infrarenal AAAs with complex aortic anatomies. This stent-graft system utilizes nitinol stent and polyester graft technology in an ultra-low profile delivery system, which assists the physician in deploying the device in a controlled, consistent, and precise manner within the aortic neck and iliac arteries. By isolating the aneurysmal sac, the system provides an alternative blood flow path to relieve pressure on the arterial vessel walls and minimize aneurysm growth and the potential for aneurysm sac rupture.

ELIGIBILITY:
1. Obtain an independent assessment by an uninvolved physician.
2. Obtain informed consent from the patient or legal representative. The consent form used should provide information pertinent to the patient's specific situation. (If appropriate, the study consent form may be used with an addendum to inform the patient of concerns specific to their situation.)
3. Obtain clearance from the institution in accordance with their policies.
4. Notify the institutional review board and comply with their procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michel S Makaroun, MD, Principal Investigator — University of Pittsburgh; Takao Ohki, MD, Principal Investigator — Jikei University School of Medicine
Locations (1):
- Cordis Corporation, Fremont, California, United States